CLINICAL TRIAL: NCT00264043
Title: Distal Protection Combined With Velocity in Coronary Arteries and SVBG Registry.
Brief Title: The Study to Evaluate Patient Outcome Using Distal Protection Combined With the BX Velocity.
Acronym: DISCOVER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll, Cordis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC99-09
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): AngioGuard™ device and Bx Velocity™ stent
  Interventions: Device: emboli capturing guidewire device combined with stent

INTERVENTIONS:
Device: emboli capturing guidewire device combined with stent — AngioGuard™ device and Bx Velocity™ stent
  Other Names: emboli capturing guidewire device; PTCA

SUMMARY:
The primary objective is to evaluate the use of the AngioGuard™ device combined with the Bx Velocity™ on patient outcome at one month.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multi-center trial. Patients will be treated with the AngioGuard™ device and Bx Velocity™ stent and will be followed for six-months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Unstable angina pectoris (Braunwald classification B & C, I-II-III, native vessels)
* or lesion located in the SVG;
* Single de novo or restenotic lesion requiring treatment in a major native coronary artery or saphenous vein graft;
* The vessel diameter to place the AngioGuard™ device in must be > 3 and < 5.5 mm (6.5 when the 7mm AngioGuard™ is available);
* Target lesion stenosis is >50% and <100% (TIMI 1).

Exclusion Criteria:

* A Q-wave or non-Q-wave myocardial infarction within the preceding 72 hours unless the CK and CK-MB enzymes are back to normal;
* More than one coronary artery is 100% occluded;
* Patient has unprotected left main coronary disease with > 50% stenosis;
* Patient has an ostial target lesion;
* Significant (>50%) untreated stenosis proximal or distal to the target lesion that will be treated during the procedure, since this may require revascularization or impede runoff;
* Ejection fraction <30%;
* Totally occluded vessel (TIMI 0 Level).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2000-05; Primary Completion 2002-02 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
clinical success of the AngioGuard™ device combined with the Bx Velocity™ stent | 1 month

SECONDARY OUTCOMES:
successful placement and retrieval without embolic occlusions of vessels distal to the position of the device | post-procedure
overall survival rates | 1 month and 6 months
device evaluation | post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Grube, MD, Principal Investigator — Herzzentrum Siegburg GMBH
Locations (1):
- Herzzentrum Siegburg GMBH, Siegburg, Germany